CLINICAL TRIAL: NCT01250093
Title: Acupuncture Compared With "Sham" Acupuncture for Treatment of Chronic Neck Myofascial Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Mei-Yuan Sun, Nantou Hospital
Other Study IDs: Nantou
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2008-10

CONDITIONS: Chronic Neck Myofascial Pain Syndrome
MeSH Terms: interventions — Acupuncture Therapy

INTERVENTIONS:
Device: acupuncture

SUMMARY:
In order to investigate the therapeutic effect of acupuncture on chronic neck myofacial pain syndrome, the investigaotrs designed a pilot study of a single-blind randomized controlled trial. A total of 34 chronic neck myofacial pain syndrome patients were selected from Department of Neurology of Nantou Hospital, Department of Health. The age ranged from 18 to 85, and all subjects were full informed consent and volunteers. They were divided into two groups of 17 subjects randomly as follows: acupuncture group, acupuncture stainless needles were inserted into bilateral Fenhchi, Jianliao and Houxi acupoints, respectively. The acupuncture needles then were manual twist and de Qi, and remain for 20 min; sham acupuncture group, the methods were identical the acupuncture group, but acupuncture stainless needles were inserted into subcutaneous tissue only. All the subjects were treated with acupuncture two times per week and continuously three weeks, i.e. Six times acupuncture treatment. The therapeutic effect of acupuncture was assessed before and finishing six times acupuncture treatment, and four weeks and twelve weeks after stopping acupuncture, respectively. The index of acupuncture therapeutic effect was according to the range of motion (ROM) of the cervical spine, the intensity of pain (Short-Form McGill Pain Questionnaire; SF-MPQ) and quality of life (SF-36). The investigators expect acupuncture apply to bilateral Fenhchi, Jianliao and Houxi acupoints may relief the pain and motion of chronic neck facial pain syndrome patient, and also improves the life quality.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 year-old patients with neck myofascial pain for more than one month; not received any treatment in the two weeks before participating this study

Exclusion Criteria:

* Fracture or surgery of the cervical spine; Cervical radiculopathy or myelopathy; Any rheumatic disorder; Systemic disorders; Major psychiatric disorder, alcoholism or substance abuse; Coagulation dysfunction, or related medicines; Pregnancy; Contraindications to acupuncture; Refused to sign consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-01 (Actual)